CLINICAL TRIAL: NCT01637662
Title: Mechanisms and Biological Markers During Headache Induced by Natriuretic Peptides
Brief Title: Natriuretic Peptide's Headache Inducing Characteristics and Effects on the Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, Danish Headache Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: H-3-2012-065
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Natriuretic Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects (Experimental)
  Interventions: Drug: Natriuretic peptides

INTERVENTIONS:
Drug: Natriuretic peptides — I.V. infusion between 0.2-3 microgram over 20 minutes

SUMMARY:
To investigate headache score and accompanying symptoms during and after infusion of the natriuretic peptides.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-40
* 50-100 kg
* Fertile women must use safe contraceptives (IUD, oral contraceptives, surgical sterilisation and long lasting gestagen.

Exclusion Criteria:

* Tension type headache more than once/month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the halflife for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Headache intensity, mean velocity of blood flow in the middle cerebral artery (VmeanMCA), superfical temporal artery diameter, PetCO2, adverse events and vital signs were recorded at T-10, T0 and then every 10 min until 120 min after start of infusion. | Every 10 min.

SECONDARY OUTCOMES:
All subjects were asked to complete a headache diary every hour until 10 h after the discharge. The diary included headache characteristics and accompanying symptoms according to the International Headache Society (IHS 2004) | 10 hours after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark